CLINICAL TRIAL: NCT06607718
Title: Hyperproteic Oral Supplementation With Vitamin D and Resistance Training in Older Patients Admitted to the Acute Unit (SERIA)
Brief Title: Nutritional and Exercise Intervention in Older Adults Admitted to the Acute Care Unit (SERIA)
Acronym: SERIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 041/23
Record Dates: First submitted 2024-09-04; First posted 2024-09-23 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Malnutrition; Protein; Older; Sarcopenia
Keywords: Oral Nutritional Supplementation; Resistance trainning; Sarcopenia; Older adults; Acute Care
MeSH Terms: conditions — Kwashiorkor; Sarcopenia | interventions — Resistance Training; Dietary Supplements; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, pragmatic study with blinded outcome measurement.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Ultrasound measurements, MNA and bioimpedance are being performed at all three visits by an investigator blinded to the assigned group. In addition, the person carrying out the data analysis will also be blinded to the assigned group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Resistance Training (RT) (Experimental): They are performing programmed physical exercise started on the day of admission, focusing on muscle strength gain, and they are being taught how to continue exercising three times a week after discharge from hospital. Lower limb strength exercises (squats and knee extensions) and upper limb strength exercises (elbow flexion, lateral and frontal raises, and tractions) were performed. A progression of the load are being made by increasing one set per month and 2 to 4 repetitions per month depending on the patient's capabilities.
  Interventions: Other: Resistance Training
- Oral Nutritional Supplementation (ONS) (Experimental): They are receiving a hypercaloric, hyperproteic, oral nutritional supplement with vitamin D and CaHMB (ß-hydroxy-ß-methylbutyrate) (Ensure Plus Advance®), at a dose of two packets per day in two or more doses for 3 months.
  Interventions: Dietary Supplement: Oral Nutritional Supplementation
- Control Group (CG) (Sham Comparator): They are being treated according to standard clinical practice, which includes information from the health professionals on the ward on recommended dietary and exercise guidelines. When the treating team considers the use of an oral nutritional supplement to be indicated, it is being prescribed.
  Interventions: Other: Control Group
- Resistance Training (RT) and Oral Nutritional Supplementation (ONS) (Experimental): They receive joint treatment
  Interventions: Other: Resistance Training; Dietary Supplement: Oral Nutritional Supplementation

INTERVENTIONS:
Other: Resistance Training — Resistance training for elderly patients in the acute care unit.
  Other Names: RT
  Arms: Resistance Training (RT); Resistance Training (RT) and Oral Nutritional Supplementation (ONS)
Dietary Supplement: Oral Nutritional Supplementation — To receive two daily packs of a hypercaloric and hyperproteic oral nutritional supplement for 3 months.
  Other Names: ONS
  Arms: Oral Nutritional Supplementation (ONS); Resistance Training (RT) and Oral Nutritional Supplementation (ONS)
Other: Control Group — No intervention
  Other Names: CG
  Arms: Control Group (CG)

SUMMARY:
This is a randomised, parallel, single-blind clinical trial. Objectives: to evaluate: the impact of the intervention on nutritional status, body composition, strength, the prevalence of sarcopenia and physical performance at discharge and three months later..

DETAILED DESCRIPTION:
Design: A randomised controlled clinical trial with four parallel groups is being conducted with older adults admitted to an acute geriatric unit at risk of malnutrition or with malnutrition. The participants are randomly assigned to one of the groups. Three assessment visits are being conducted: at admission, discharge, and three months later.

Setting: The study is being conducted in the Unidad de Agudos del Servicio de Geriatría at Hospital Universitario Ramón y Cajal, by the Servicio Madrileño de Salud (SERMAS).

Interventions: four groups: 1) a resistance training group (RT); 2) an oral nutritional supplementation group (ONS); 3) a combination of RT and ONS (RT+ONS); and a control group (CG). The patients in the RT group follow individualized RT sessions with a physiotherapist daily during the hospitalization and three weekly home sessions on their own after discharge. The sessions are structured according to the recommendations of the American College of Sports Medicine (ACSM), mainly RT.

Study population: A study of malnourished or at-risk outpatients in our setting was used to calculate the sample size. In that study, with an alpha error of 0.05 and a beta of 0.80, the minimum sample size was 14 participants per group. Our objective is to include, at least, 21 participants per group, resulting in a total of 84 participants.

Sociodemographic and clinical variables are being collected (e.g., age, sex, living situation, number of drugs, falls). Information about nutritional and functional status (e.g., MNA, gait speed, Barthel, Lawton, and FAC), body composition (e.g., weight, height, body mass index, appendicular muscle mass index measured by bioimpedanciometry (BIA)), ultrasound measurements of the anterior rectus (area, thickness, and penation angle), and muscle strength (hand grip test) is also collected.

The first descriptive analysis of the variables will include frequencies and percentages for categorical variables and means and standard deviations for continuous variables. Changes in nutritional status will be analysed as well as the interaction between nutrition and exercise by repeated measures ANOVA. The prevalence of sarcopenia and the influence of each component of the sarcopenia definition on physical performance, ADLs, emergency room visits, and new admissions. Additionally, a survival analysis will be performed to compare the four groups. To assess the quality of ultrasound measurement, the relationship between each ultrasound variable and the bioimpedance score, as well as the diagnostic criteria for malnutrition and sarcopenia, will be analysed. Furthermore, ultrasound measurements will be correlated with the estimation of muscle mass using bioimpedance analysis. A p-value less than 0.05 will be considered statistically significant.

The study is being conducted under the ethical standards set forth by the Comité de Ética de Investigación con Medicamentos (CEIm) of the Hospital Universitario Ramón y Cajal. Each participant is informed about the study and signs the informed consent before inclusion. The study has been designed and subsequently evaluated under Law 14/2007 on Biomedical Research, the ethical principles of the Declaration of Helsinki of the World Medical Association on Ethical Principles for Medical Research on Human Beings, as well as the other ethical principles and legal regulations applicable according to the characteristics of the study.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the Unidad de Agudos (Geriatric Acute Care) del Servicio de Geriatría at HU Ramón y Cajal who are at risk of malnutrition or malnutrition (defined with a MNA-SF score ≤ 11) and who sign the informed consent form.

Exclusion Criteria:

* patients with estimated discharge within 72 hours.
* Re-admissions (defined as previous admission in the Geriatric Acute Care in the last 3 months)
* Patients taking ONS for more than two weeks.at the time of admission.
* Patients suffering any illness or condition that prevents or contraindicates resistance physical exercise. and oral food intake.
* Food allergies or intolerances that contraindicate the SNO.
* Patients with advanced dementia (GDS stage 7) or palliative care.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Mini Nutritional Assessment (MNA) | 12 weeks
  Screening tool to help identify malnourished elderly people or those at risk of malnutrition on a scale of 0 to 30. The higher the value, the better the nutritional status of the older adult.

SECONDARY OUTCOMES:
Hand grip test | 12 weeks
  Measurement of hand grip strength using a hand-held dynamometer.
Body Mass Index (BMI) | 12 weeks
  Is a mathematical ratio that associates the mass and the size of an individual BMI = weight / height ^2
Appendicular Skeletal Muscle mass Index (ASMI) | 12 weeks
  It is the sum of muscle masses of the four limbs measured with BIA.
4-m-test | 12 weeks
  It consists of assessing the patient's usual walking speed over a distance of 4 metres.
Barthel's index | 12 weeks
  Test to assess the patient's ability to perform basic activities of daily living on a scale of 0 to 100. The higher the value, the greater the independence of the older adult.
Lawton-Brody scale | 12 weeks
  Test to assess the patient's ability to perform instrumental activities of daily living on a scale of 0 to 8. The higher the score, the greater the functional capacity of the older adult.
Functional Ambulation Classification (FAC) | 12 weeks
  Test to assess a person's ability to walk with a score from 0 to 5. The higher the score, the greater the walking independence.
Cross-sectional area | 12 weeks
  An ultrasound is performed in the middle of the anterior rectus, measuring from the patella to the anteroinferior iliac spine. Through a cross section the image is frozen and the area of the volume of the anterior rectum at that point is traced. The area is noted in cm^2.
Thickness | 12 weeks
  An ultrasound is performed in the middle of the anterior rectus, measuring from the patella to the anteroinferior iliac spine. Through a cross section the image is frozen and a straight line of the thickness of the center of the anterior rectus is drawn at that point. The distance is noted in mm.
Penile angle of a muscle | 12 weeks
  An ultrasound is performed in the middle of the anterior rectus, measuring from the patella to the anteroinferior iliac spine. Unlike the other measurements, the ultrasound image is taken in the longitudinal section. The penile angle of a muscle is the orientation of the muscle fibers in relation to the connective tissue/tendon. It is taken by fixing one side of the angle on the connective tissue and the other side on the orientation of the muscle fibers. The value is noted in degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Montero-Errasquín, Dra., Principal Investigator — Hospital Ramon y Cajal.
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
No personal information will be shared. At the time of enrolment, each participant will be given a code. The full database of outcome variables will also not be shared.